CLINICAL TRIAL: NCT01518530
Title: Tailored Computerized Mobilization of the Cervical Spine Utilizing the Occiflex Device for the Treatment of Chronic Neck Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0086-11-HYMC
Record Dates: First submitted 2011-12-20; First posted 2012-01-26 (Estimated); Results first posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-08

CONDITIONS: Neck Pain
Keywords: Chronic Neck Pain, Occiflex, Computerized Mobilization
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Passive Mobilization Cervical Spine (Experimental): Patients with chronic neck pain according to the International Association of the Study of Pain criteria of the following types: facet joint disorder, post-whiplash injury, myofascial pain syndrome.
  Interventions: Device: Occiflex Robotic Intervention System

INTERVENTIONS:
Device: Occiflex Robotic Intervention System — Occiflex is a robotic system which is comprised of a cradle moved in a three dimension space with six degrees of freedom. It allows the therapist to tailor a personalized course of 3-D mobilization of the head and neck.

SUMMARY:
The study is intended to examine the safety and efficacy of computerized mobilization of the neck for the treatment of patients with chronic neck pain. This is a third continuation study aimed at examining the Occiflex Robotic System. This time we will be studying tailored or personalized three dimensional movement of the neck.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic neck pain: post-whiplash injury, myofacial pain, cervical facet joint disease and idiopathic chronic neck pain

Exclusion Criteria:

* Patients with cervical radiculopathy Myelopathy Discopathy Malignancy involving the neck or cervical spine Severe Osteoporosis Severe skin disorder Psychiatric disorders Cervical disc herniation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2012 to February 2012 twenty-three patients were screened and 10 were found to be eligible in the Physical Therapy Department of the Hillel Yaffe Medical Center.
Pre-assignment Details: One recruited patient was dropped because of protocol violation.
Groups:
- Chronic Neck Pain Patients Treated With Occiflex: Occiflex is a computerized robotic system for the accurate 3-dimensional mobilization of the head and neck.
Period: Active Treatment Period
Arm/Group | Chronic Neck Pain Patients Treated With Occiflex
Started | 10
Completed | 9
Not Completed | 1
Period: Post-Treatment Follow-up
Arm/Group | Chronic Neck Pain Patients Treated With Occiflex
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: One patient dropped out of the experiment due to lack of necessary documentation required for inclusion.
Groups:
- Patients With Chronic Neck Pain Treated With Occiflex: Occiflex is a computerized robotic system for the accurate 3-dimensional mobilization of the head and neck.
Arm/Group | Patients With Chronic Neck Pain Treated With Occiflex
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Region of Enrollment [Number; unit: participants]
  Israel | 10

OUTCOME MEASURES:

1. Primary Outcome: Occiflex Device Safety
Description: A meticulous documentation of any serious adverse effect will be made. Any minor side effects will be recorded with an emphasis on the possible relationship to the treatment. The number of minor and serious adverse effects out of 360 therapeutic sessions will be noted.
Time Frame: 6 weeks
Measure: Number; unit: Number of adverse effects
Arm/Group | Patients With Chronic Neck Pain Treated With Occiflex
Number analyzed (Participants) | 9
Number of adverse effects | 26

2. Secondary Outcome: Efficacy as Per the NDI-Neck Disability Index
Description: The most important instrument used to measure efficacy of treatment in patients with chronic neck pain will be used. A score of 0-50, where 50 denotes maximal disability due to chronic neck pain will be documented.
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Patients With Chronic Neck Pain Treated With Occiflex
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 7/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Chronic Neck Pain Treated With Occiflex (N=9)
Headache (Nervous system disorders) | 4 (8)
Dizziness (Ear and labyrinth disorders) | 4 (8)
Neck Pain (Musculoskeletal and connective tissue disorders) | 5 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No